CLINICAL TRIAL: NCT07202507
Title: Proof-of-Concept Study of the SNOEZELEN Device on Anxiety Symptoms in Patients Hospitalized for Chemotherapy in a Pediatric Oncology Department
Acronym: SNOOZE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: PETRARQUE (Unknown); Scalab CNRS 9193 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SNOOZE-2501; 2025-A00760-49 (Other: ANSM)
Record Dates: First submitted 2025-07-01; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Snoezelen; Pediatric Cancer; Symptomatologie Anxieuse; Chimiothérapie
Keywords: Snoezelen; Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Snoezelen (Experimental): Participants will be enrolled between their first chemotherapy cycle (without Snoezelen) and their second cycle (with Snoezelen). During the study, they will complete self-report questionnaires assessing anxiety, depression, quality of life, and nausea. They will receive 45-minute Snoezelen sessions every two days during their second hospitalization. After the final session, participants will take part in a semi-structured interview. In addition, data will be collected on medications administered (anxiolytics and antiemetics) and on the frequency of vomiting during both hospital stays.
  Interventions: Other: self-report questionnaires, research interviews

INTERVENTIONS:
Other: self-report questionnaires, research interviews — self-report questionnaires and research interviews

SUMMARY:
The goal of this clinical trial is to evaluate whether the Snoezelen multisensory relaxation approach can reduce anxiety symptoms in children and adolescents aged 8 to 17 years hospitalized for chemotherapy in a pediatric oncology unit.

Researchers will compare patients' symptoms during a chemotherapy cycle with Snoezelen sessions to a previous cycle without Snoezelen, in order to assess changes in psychological and physical well-being.

Participants will:

* Be enrolled between their first (without Snoezelen) and second (with Snoezelen) chemotherapy cycles
* Complete self-report questionnaires on anxiety, depression, quality of life, and nausea
* Receive 45-minute Snoezelen sessions every two days during their second hospitalization
* Participate in a semi-structured interview after the final session
* Provide data on medications (anxiolytics, antiemetics) and vomiting frequency during both hospitalizations

DETAILED DESCRIPTION:
This is a monocentric proof-of-concept study using mixed methods (quantitative questionnaires and qualitative interviews) to explore the potential benefits of Snoezelen as a supportive care intervention in pediatric oncology.

The goal of this interventional study (minimal risk clinical trial - RIPH2) is to evaluate the effect of the Snoezelen multisensory relaxation approach on anxiety symptoms in children and adolescents aged 8 to 17 years who are hospitalized for chemotherapy in a pediatric oncology unit.

The primary research question is:

- Does the use of Snoezelen reduce anxiety symptoms during hospitalization for chemotherapy in pediatric cancer patients?

Secondary research questions include:

* Does Snoezelen improve quality of life and reduce depressive symptoms?
* Does Snoezelen reduce nausea and vomiting during chemotherapy? Researchers will compare participants' symptoms before and after a chemotherapy cycle with Snoezelen sessions, and contrast these with data from the previous cycle without Snoezelen.

Participants will:

* Be enrolled between their first (without Snoezelen) and second (with Snoezelen) chemotherapy cycles
* Complete self-report questionnaires assessing anxiety (GAD-7, SCARED), depression (CDI), quality of life (PedsQL), and nausea (BARF scale)
* Receive 45-minute Snoezelen sessions every two days during their second hospitalization for chemotherapy
* Participate in a semi-structured research interview after the final Snoezelen session The study will also collect data on medications administered (anxiolytics, antiemetics) and the frequency of vomiting episodes during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* New patient
* Treated in the Paediatrics/AJA department of the Oscar Lambret Centre for cancer (all types of cancer)
* Hospitalisation for several days
* Highly emetogenic chemotherapy treatment: this corresponds to all in-patient treatments carried out in the Paediatrics/AJA department.
* Age at diagnosis : ≥ 8 years and < 18 years.
* French language
* Information for the patient and those with parental authority; consent signed by the patient and those with parental authority.
* Valid social security cover

Exclusion Criteria:

* Contraindication to SNOEZELEN:

  * Claustrophobia
  * Presence of psychiatric, addictive or cognitive disorders that would prevent compliance with the protocol requirements;
* State of health not allowing participation in the study (severe fatigue, symptoms refractory to treatment).
* Pregnant or breast-feeding women

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Semi-structured research interview | At the end of the 2nd course of chemotherapy and no more than 2 weeks after the last Snoezelen session, 1 month after inclusion
  Interview with a research psychologist to find out how teenage children feel

SECONDARY OUTCOMES:
Generalized Anxiety Disorder - GAD-7 | Before the 2nd chemotherapy treatment, before the 1st Snoezelen session and At the end of the 2nd chemotherapy treatment and no more than 2 weeks after the last Snoezelen session = at 15 days and at 1 months
  Self-questionnaire
Anti-emetic treatments | Periprocedural
  Collection of anti-emetic treatments administered during hospitalisation
Child-Self Report - PedsQL | Before the 2nd chemotherapy treatment, before the 1st Snoezelen session and At the end of the 2nd chemotherapy treatment and no more than 2 weeks after the last Snoezelen session = at 15 days and at 1 months
  Self-questionnaire (ages 8-12 or 13-18)
Number of vomits | Periprocedural
  Collection of the number of vomits during hospitalisation
Anxiolytic treatments | Periprocedural
  Collection of anxiolytic treatments received during hospitalization
BARF scale (Baxter Retching Faces) | Before the 2nd chemotherapy treatment, before the 1st Snoezelen session and At the end of the 2nd chemotherapy treatment and no more than 2 weeks after the last Snoezelen session = at 15 days and at 1 months
  Evaluation of nausea/vomiting
Children's Depression Inventory - CDI | Before the 2nd chemotherapy treatment, before the 1st Snoezelen session and At the end of the 2nd chemotherapy treatment and no more than 2 weeks after the last Snoezelen session = at 15 days and at 1 months
  Self-questionnaire
Child Anxiety Related Emotional Disorders - SCARED | Before the 2nd chemotherapy treatment, before the 1st Snoezelen session and At the end of the 2nd chemotherapy treatment and no more than 2 weeks after the last Snoezelen session = at 15 days and at 1 months
  Self-questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No